CLINICAL TRIAL: NCT03726021
Title: Clinical Study of Irinotecan,Oxaliplatin, and S1 in Patients With Advanced Pancreatic Cancer
Brief Title: Study of Irinotecan,Oxaliplatin, and S1 in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2018-10-28
Record Dates: First submitted 2018-10-27; First posted 2018-10-31 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Overall Survival
Keywords: overall survival; Irinotecan; Oxaliplatin; S1; Chemotherapy
MeSH Terms: interventions — Irinotecan; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Experimental: Irinotecan,Oxaliplatin, and S1
  * S1 will be administered orally days 1 and 14 of a 21 day cycle
  * Irrinotecan 165 mg/m2 and Oxaliplatin 85mg/m2 will be administered IV days 1 of a 21 day cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Treatment consists of treatment with Irinotecan 165mg/m2, Oxaliplatin 85mg/m2 on day 1, and S1 40mg orally on day 1-14, every 21 days each cycle. Treatment will be administered until untolerable toxicities or progression or subject death, or either the subject or sponsor discontinues the study.
  Interventions: Drug: Irinotecan,Oxaliplatin, and S1

INTERVENTIONS:
Drug: Irinotecan,Oxaliplatin, and S1 — Drug: Irinotecan is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells.
  Drug: Oxalipatin Oxaliplatin is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells
  Drug: S1 is a chemotherapy agent. Chemotherapy agents are medicines that kill cancer cells
  Other Names: CPT-11/L-OHP/TS-1

SUMMARY:
To identify the efficiency of Irinotecan, Oxaliplatin, and S1 in patients with previously untreated local regional or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This research study is a Phase 2 clinical trial. It will test the efficiency and safety of an investigational drug f Irinotecan,Oxaliplatin, and S1, with the goal of determining the OS of advanced pancreatic adenocarcinoma..

Subjects must have a newly diagnosed stage 4 untreated metastatic pancreatic ductal cancer and meet all inclusion/exclusion criteria.

Treatment consists of treatment with Irinotecan 165mg/m2, Oxaliplatin 85mg/m2 on day 1, and S1 40mg orally on day 1-14, every 21 days each cycle. Treatment will be administered until untolerable toxicities or progression or subject death, or either the subject or sponsor discontinues the study.

ELIGIBILITY:
Inclusion Criteria:

* • Cytologically- or histologically-confirmed pancreatic adenocarcinoma or poorly differentiated pancreatic carcinoma that is metastatic to distant sites.

  * Other histologies such as neuroendocrine and acinar cell carcinoma are excluded.
  * No prior chemotherapy for locally advanced or metastatic pancreatic cancer.
  * Patients are eligible if they received adjuvant treatment after surgical resection
  * Participants are required to have measurable disease (RECIST v1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan. See section 11 for the evaluation of measurable disease.
  * Participants enrolled must have disease that is accessible for tumor biopsies and must agree to a pre-treatment tumor biopsy.
  * Age ≥ 18 years. Because no dosing or adverse event data are currently available in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
  * ECOG performance status ≤2 (see Appendix A)
  * Patients must have completed any major surgery or open biopsy ≥4 weeks from start of treatment.
  * Participants must have adequate organ and marrow function as defined below:

    * Absolute neutrophil count ≥1,500/mcL
    * Platelets ≥100,000/mcL
    * Total bilirubin ≤1.5 × institutional upper limit of normal
    * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
    * Creatinine ≤1.5 × institutional upper limit of normal OR
    * Creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × upper limit of normal.
  * Negative serum pregnancy test for women of childbearing potential.
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* • Prior chemotherapy or any other investigational agents for the treatment of locally advanced or metastatic pancreatic cancer

  * Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents.
  * Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Screening for brain metastases with head imaging is not required.
  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to above drugs or other agents used in study.
  * History of prior or current synchronous malignancy, except:

    o Malignancy that was treated with curative intent and for which there has been no known active disease for >3 years prior to enrollment
  * Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, NYHA class III/IV congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The overall survival in this population of patients. | Time Frame: 2 years
  The overall survival of the enrolled patients from start the combination treatment of Irinotecan, Oxaliplatin, and S1.

SECONDARY OUTCOMES:
The response rate in this population of patients. | Time Frame: 2 years
  Number of participants with clinical response assessed by RECIST 1.1 criteria on imaging every 4 weeks with the combination of Irinotecan,Oxaliplatin, and S1.
The progression free survival in this population of patients. | Time Frame: 2 years
  The progression free survival of the enrolled patients from start the combination treatment with Irinotecan,Oxaliplatin, and S1.
The toxicities in this population patients | Time Frame: 2 years
  Adverse events were recorded and classified from start the treatment by grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: youxin ji, MD, Principal Investigator — Qingdao Central Hospital
Locations (1):
- Qingdao Central Hospital, Qingdao, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nie K, Zhang L, You Y, Li H, Guo X, Zhang Z, Zhang C, Ji Y. Irinotecan combined with oxaliplatin and S-1 in patients with metastatic pancreatic adenocarcinoma: a single-arm, three-centre, prospective study. Ther Adv Med Oncol. 2020 Nov 12;12:1758835920970843. doi: 10.1177/1758835920970843. eCollection 2020. PMID 33240399